CLINICAL TRIAL: NCT00074542
Title: A Phase III Randomized, Placebo-Controlled, Double-Blind, Parallel Group, Multi-Centre Study to Assess the Efficacy and Safety of Omega-3 Free Fatty Acids (Epanova™) for the Maintenance of Symptomatic Remission in Subjects With Crohn's Disease
Brief Title: An Efficacy and Safety Study of Omega-3 Free Fatty Acids (Epanova™) for the Maintenance of Symptomatic Remission in Subjects With Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tillotts Pharma AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol TP0308 (EPIC-2)
Record Dates: First submitted 2003-12-15; First posted 2003-12-16 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2005-10

CONDITIONS: Crohn's Disease
Keywords: Crohn's; colon; small bowel; inflammation; steroid therapy; free fatty acids
MeSH Terms: conditions — Crohn Disease; Inflammation

INTERVENTIONS:
Drug: Epanova™ (Omega-3 Free Fatty Acids)

SUMMARY:
The purpose of this study is to see if Epanova™ is able to maintain the symptomatic remission in subjects with Crohn's Disease who are responding to steroid induction therapy.

Patient safety and quality of life will also be monitored throughout the study.

DETAILED DESCRIPTION:
Crohn's disease is a chronic inflammatory disorder that frequently involves the colon and small bowel. Patients commonly experience abdominal pain, diarrhea, and malaise which result in decreased quality of life and an increased risk of chronic disability and unemployment.

Currently available therapeutic options for the maintenance of remission in Crohn's disease are inadequate. Patients' quality of life is often severely diminished. A clear need exists for well-tolerated drugs that can reliably reduce the risk of a disease relapse.

In recent years considerable attention has been focused on dietary marine fish oils as a means of treating several chronic inflammatory disorders including Crohn's disease. Fish oils have been found to reduce the inflammation and the severity of lesions in animal models of inflammatory bowel disease.

Commercially available fish oils are supplied as fatty acid triglycerides or ethyl esters and are often associated with unpleasant side effects such as nausea, flatulence, diarrhea and belching. These adverse effects limit administration of high doses of these preparations. Several studies have demonstrated the superior absorption across intestinal membranes of free fatty acids in comparison with triglycerides and ethyl esters. Epanova™ is being developed as a well-tolerated means of delivering a high concentration of marine fish oils as free fatty acids. Additionally, the gelatin coating of the capsules consists of a permeable polymer that results in a delayed release of the active compounds thus reducing the frequency of adverse events.

The objectives of this clinical trial are as follows:

Primary Objective:

* To assess the ability of Epanova™ to maintain symptomatic remission in subjects with Crohn's Disease who are responding to steroid induction therapy

Secondary objectives:

* To assess the safety and tolerability of Epanova™
* To assess the ability of Epanova™ to maintain the quality of life in subjects with Crohn's Disease who are responding to steroid induction therapy
* To assess the efficacy of Epanova™ by Crohn's Disease Activity Index (CDAI), Investigator and Subject Global Ratings, employment status and use of Crohn's Disease related medical visits in subjects with Crohn's Disease who are responding to steroid induction therapy

ELIGIBILITY:
Key Inclusion Criteria:

* symptomatic active Crohn's disease (requiring a 16-week course of induction steroid therapy at a starting dose of prednisone 40 mg or budesonide 9 mg daily)
* respond to induction therapy (CDAI<150) following 8 weeks of steroid tapering regimen to prednisone 20 mg or budesonide 6 mg daily
* Crohn's disease of at least 3 months duration
* 16 years of age or older

Key Exclusion Criteria:

* intolerance of omega-3 free fatty acid (FFA)
* intolerance of both prednisone and budesonide
* ongoing therapy for Crohn's disease with: 5-ASA compounds, immune modifiers, systemic antibiotics, tube feeding
* received in the past 3 months: systemic steroid therapy (other than study prednisone or budesonide induction therapy), azathioprine, 6-mercaptopurine, methotrexate, cyclosporine, probiotic products, preparations containing omega-3 fatty acids
* received in the past 6 months: biologicals e.g. enbrel, infliximab, monoclonal antibody, mycophenolate, tacrolimus, thalidomide, other immune modifiers and/or investigational products
* chronic narcotic analgesics for pain control
* short bowel syndrome, ostomy or need for bowel surgery for Crohn's disease, bowel obstruction or resection in the past 3 months
* malignancy, clinically significant impairment or conditions which could interfere with the evaluation of the trial medication
* clinically relevant hematology, liver and renal function laboratory tests
* known allergy to fish or fish products

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 364
Dates: Start 2002-09; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (31):
- United States (10):
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Northwestern University Medical School, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Carle Clinic Association, Urbana, Illinois
  - University of Louisville, Department of Surgery, Louisville, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Gastroenterology Specialties, P.C., Lincoln, Nebraska
  - Long Island Clinical Research Associates, Great Neck, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
- Canada (21):
  - Health Sciences Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Victoria General Hospital, Halifax, Nova Scotia
  - London Health Sciences Centre (South Street Campus), London, Ontario
  - London Health Sciences Centre (University Campus), London, Ontario
  - The Ottawa Hospital (Civic Campus), Ottawa, Ontario
  - Sunnybrook & Women's College HSC, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - CHUQ - Pavillon St-François d'Assise, Montreal, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hôpital Saint-Luc, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHUQ-Hôtel-Dieu de Québec, Québec, Quebec
  - Hôpital St-Sacrement, Québec, Quebec

REFERENCES:
- [Background] Belluzzi A, Brignola C, Campieri M, Pera A, Boschi S, Miglioli M. Effect of an enteric-coated fish-oil preparation on relapses in Crohn's disease. N Engl J Med. 1996 Jun 13;334(24):1557-60. doi: 10.1056/NEJM199606133342401. PMID 8628335
- [Derived] Feagan BG, Sandborn WJ, Mittmann U, Bar-Meir S, D'Haens G, Bradette M, Cohen A, Dallaire C, Ponich TP, McDonald JW, Hebuterne X, Pare P, Klvana P, Niv Y, Ardizzone S, Alexeeva O, Rostom A, Kiudelis G, Spleiss J, Gilgen D, Vandervoort MK, Wong CJ, Zou GY, Donner A, Rutgeerts P. Omega-3 free fatty acids for the maintenance of remission in Crohn disease: the EPIC Randomized Controlled Trials. JAMA. 2008 Apr 9;299(14):1690-7. doi: 10.1001/jama.299.14.1690. PMID 18398081
- See also: Sponsor's Website — http://www.tillotts.com